### **PROTOCOL**

| Transbronchial needle aspiration with cryobiopsy in the diagnosis of mediastinal disease: a randomised trial |
|---|
| 2.1 |
| NCT04572984 |
| Professor Felix JF, Department of<br>Pneumology and Critical Care Medicine,<br>Thoraxklinik, and Translational Lung<br>Research Center Heidelberg, University<br>of Heidelberg, Heidelberg, Germany |
| Ye Fan, Department of Respiratory<br>Disease, Xinqiao Hospital, Third Military<br>Medical University, Chongqing, China |
| University of Heidelberg, Heidelberg,<br>Germany<br>Xinqiao Hospital, Third Military Medical<br>University, Chongqing, China |

**Chief Investigator Signature:** 

# **Confidentiality Statement**

Felix Holl

This document contains confidential information that must not be disclosed to anyone other than the Sponsor, the Investigator Team, HRA, host organisation, and members of the Research Ethics Committee and Regulatory Authorities unless authorised to do so.

# **TABLE OF CONTENTS**

| 1. E | Background | 1 |
|------|-----------------------------------------------------------|----|
| 2. ( | Objective | 1 |
| 3. 7 | Frial design and procedure | 1 |
| | 3.1 Trial Participants | 2 |
| | 3.2 Sample size | 3 |
| | 3.3 Randomisation and blinding | 3 |
| | 3.4 Patient withdrawal | 4 |
| 4. ٦ | Frial interventions | 4 |
| | 4.1 Sedation | 4 |
| | 4.2 EBUS procedure | 5 |
| | 4.3 EBUS-TBNA | 6 |
| | 4.4 Transbronchial mediastinal cryobiopsy after EBUS-TBNA | 6 |
| | 4.5 Postbiopsy | 7 |
| | 4.6 Procedure interruption | 7 |
| | 4.7 Histological assessment | 8 |
| | 4.8 Patient follow-up | 8 |
| 5. 8 | Study endpoints | 9 |
| 6. [ | Data analysis | 9 |
| 7. E | Ethical considerations | 10 |
| 8. F | Risks and benefits | 10 |
| 9. F | Privacy and personal information protection | 11 |
| 10. | Funding | 11 |
| 11 | Reference | 11 |

1. Background

Mediastinal and hilar lymphadenopathy can be manifested in both malignant and benign

disorders. Accurate timely diagnosis of mediastinal disease is essential for choosing

appropriate treatment and for predicting prognosis, which usually requires sufficient samples

qualified for pathological and molecular assessment. Endobronchial ultrasound-guided

transbronchial needle aspiration (EBUS-TBNA) is a minimally invasive and safe technique

that is widely employed for the sampling of mediastinal lesions<sup>1</sup>. Clinical guidelines

recommended that EBUS-TBNA is a preferred and initial modality for the invasive staging of

non-small cell lung cancer (NSCLC)<sup>2, 3</sup>. However, the relatively limited amount of intact tissue

obtained might restrict its diagnostic yield in mediastinal diseases of other etiologies<sup>4, 5</sup>.

We recently demonstrated that transbronchial mediastinal cryobiopsy provides larger

amounts of intact tissue and improves the overall diagnostic yield as compared to

EBUS-TBNA<sup>6, 7</sup>. The excellent performance of this approach, particularly in non-lung cancer

diseases, suggests a potentially additive value of mediastinal cryobiopsy to the standard

sampling strategy<sup>7</sup>.

2. Objective

We aim to prospectively evaluate the diagnostic accuracy and the safety of adding

transbronchial mediastinal cryobiopsy to standard sampling in mediastinal diseases.

3. Trial design and procedure

This is a prospective, mutlicentre, randomised, comparative, diagnostic accuracy study,

which is designed to evaluate diagnostic value and safety of combined application of

EBUS-TBNA and mediastinal cryobiopsy. The study is designed and reported following the

Consolidated Standards for Reporting Trials (CONSORT).

Date and version No: 8th February 2022 version 2.1

3.1 Trial Participants

Consecutive individuals who need bronchoscopic diagnosis based on suspicion of either

benign or malignant disease in mediastinal or hilar lymph nodes or masses, and who have

completed preoperative examinations, are prospectively enrolled by the team member from

each of the participating centres according to the inclusion criteria. Those individuals not

suitable for bronchoscopy or mediastinal biopsy or who meet the exclusive criteria are

excluded from study. The details of the inclusive and exclusive criteria are presented below.

3.1.1 Inclusive criteria

Aged ≥ 15 years old;

Patients with at least one mediastinal lesion with a short-axis ≥ 1 cm that is detected by

thoracic image;

Patients with recently discovered mediastinal lesions, clinical respiratory symptoms of

cough, expectoration, thoracalgia, apnea, or complicated lung lesions implicated by thoracic

image, which indicates a need for biopsy to identify the underlying etiology;

Patients should have undergone necessary preoperative laboratory examinations and

other examinations such as cardiac ultrasound or CTA when necessary, in order to exclude

potential contradictions;

Patient is willing and able to give informed consent for participation in the study.

3.1.2 Exclusive criteria

Patients with contradictions to endoscopic examination, such as severe cardiopulmonary

diseases, coagulation disorders, intolerance to anesthesia or endoscopic operation,

psychiatric disorders, or severe neurosis, and so on;

The EBUS procedure fails to detect the mediastinal lesion;

The mediastinal lesions are actually cysts or abscess:

Patients need for additional procedures other than EBUS examination (such as

2

endobronchial biopsy);

Patients could not provide full informed consent;

Patients have been previously randomised to an arm of the present trial or involved in other clinical trials in the recent 3 months;

Patients have any other conditions that are considered to be inappropriate to be involved in this study.

# 3.2 Sample size

Sample size of this study is calculated by Power Analysis version 11.0 and Sample Size version 11.0 software using two independent proportions analysis.

#### Two Independent Proportions (Null Case) Power Analysis

Numeric Results of Tests Based on the Ratio: P1 / P2

H0: P1/P2=1. H1: P1/P2=R1<>1. Test Statistic: Z test with pooled variance

| | Sample<br>Size | The second secon | Prop H1<br>Grp 1 or | Prop<br>Grp 2 or | Ratio | Ratio | | | |
|---|---|---|---|---|---|---|---|---|---|
| Power | Grp 1<br>N1 | Grp 2<br>N2 | Trtmnt | Control<br>P2 | if H0<br>R0 | if H1<br>R1 | Target<br>Alpha | Actual<br>Alpha | Beta |
| 0.9015 | 130 | 2000 | 0.9348 | 0.7990 | 1.000 | 1.170 | 0.0500 | Alpha | 0.0985 |

Note: exact results based on the binomial were only calculated when both N1 and N2 were less than 100.

Sample size estimation is conducted according to the findings of our prior transbronchial mediastinal biopsy report indicating the similarly low operational risks of EBUS-TBNA and cryobiopsy (no serious adverse events have been observed in both groups), and thus the number of the required cases is calculated mainly on the basis of potential diagnosis benefit<sup>7</sup>. Assuming that the increase in the overall diagnostic yield by the combined approach is 13.5% (a threshold of 79.9%),  $\alpha$ =0.05,  $\beta$ =0.1, power is 0.9, N is calculated to be 130 for each group. The result report is presented above.

# 3.3 Randomisation and blinding

Patients will be randomised using a computer-generated blocked randomisation scheme (block size four based on a random table from an independent statistician who has no further

involvement in the actual clinical study). The allocation is stratified at the centre level. Once

study participants are deemed eligible, a member of the trial team will randomise the

participant. The random allocation sequence will not be disclosed to patients and consenting

investigators until the interventions are assigned. Because of the nature of the intervention,

neither patients nor study personnel could be masked to group assignment. The radiologists

and the pathologists are unaware of the patient recruitment for a clinical trial. The

paper-based case forms are applied to record study data, and important information such as

patient-related information and the diagnostic results, are also recorded in an electronic

system. The data are further collected by an independent research assistant. Data monitoring

is conducted at each of the centres on the basis of the the local ethic committee

recommendation.

3.4 Patient withdrawal

All patients reserve the right to withdraw from the study at any time. For those who lack

appropriate decision-making ability, the expression of dissent in any form will be taken as an

indication that they do not wish to be included and these individuals are then withdrawn.

4. Trial interventions

All the procedures are performed by the same experienced bronchoscopist from each

centre.

4.1 Sedation

Patients are in supine position. The upper airway topical anesthesia is achieved by 2%

lidocaine, and conscious sedation is achieved by intravenous injection of midazolam and

fentanyl. Oxygen is initially administrated at 1-2 L/min and increased when oxygen saturation

is lower than 90%. Patients' vital signs and pulse blood oxygen saturation are continuously

monitored.

Date and version No: 8th February 2022 version 2.1

## 4.2 EBUS procedure

In our procedure, rigid bronchoscopy is not used. An EBUS bronchoscope (BF-UC260F-OL8 or BF-UC260F, Olympus, Tokyo, Japan) is inserted into the trachea through the nose (if the nasal airway is too narrow for the EBUS bronchoscope to pass through or there are other contradictions, the oral way can be the alternative option). As the EBUS bronchoscope has been inserted in, the glottis, the trachea, the bronchuses are probed in turn. After the examination of the airway, the EBUS bronchoscope is then contacted with the airway wall, and a systematic examination of all mediastinal and hilar lymph node stations is sequentially performed according to the Mountain-Dressler lymph node map. For each lesion, the blood supply is identified by the Doppler Ultrasound and the size is measured by its long axis and short axis. The most suspicious target (lesion with disease characteristics implicated by imaging data [such as significantly enlarged size, contrast enchantment on CT imaging, high FDG uptake on PET/CT imaging, et al.]) with relatively less biopsy risk is chosen for biopsy sampling. The ultrasonic detection duration is defined as the time interval from the insertion of the bronchoscope into the nose or mouth to the moment when the mediastinal lesion is detected.

After the target is localized, EBUS-TBNA (step 4.3) with or without transbronchial mediastinal cryobiopsy (step 4.4) is performed according to the randomised group. To avoid the risk of severe bleeding, the vascularization status of the lesion is assessed by Doppler-mode blood flow imaging as previously described by Nakakima and coworkers<sup>8, 9</sup>. Lesions are classified as follows: grade 0: no blood flow or small amounts of flow; grade I: a few main vessels running toward the center of the lesion; grade II: a few punctiform or rod-shaped flow signals, a few small vessels found as a long strip of a curve; and grade III: rich flow, more than four vessels found with different diameters and a twist or helical-flow signal. If the lesion is too abundant in blood supply (Grade III), too close to large vessels, or other conditions detected by EBUS that indicates high risk of biopsy, another appropriate lesion would be considered for sampling.

#### 4.3 EBUS-TBNA

4.3.1 As the target lesion has been visualized by ultrasound, a dedicated TBNA needle (21-gauge or 22-gauge, NA-201SX-4021 or NA-201SX-4022, Olympus, Tokyo, Japan, which are the standard biopsy instruments for EBUS-TBNA as recommended by the current guideline) is passed through the working channel of the EBUS bronchoscope, and advanced through the tracheobronchial wall into the lesion under real-time ultrasound visualization, avoiding areas with abundant blood supply or massive necrosis<sup>10</sup>. After the central stylet has been removed, the suction is applied using a syringe while the needle is manipulated back and forth for 25 times within the lesion. The specimen collected in the lumen of the needle is pushed out using the central stylet and then blown by air with a syringe onto a glass slide. The specimen on the glass slide is smeared and fixed in 95% alcohol for cytologic examination. The visible tissue fragment on the glass slide and the residual specimen in the lumen of the needle are collected and transferred into the containers filled with formalin for cell block analysis. Both cell block analyses and glass slide-based cytology analyses are performed.

4.3.2 Repeat 4.3.1 for 4 times. The operation duration for TBNA is recorded from the insertion of the needle into the bronchoscope to its final exit from the working channel. Patients assigned to the combined group will receive one-time mediastinal cryobiopsy after the completion of EBUS-TBNA, which is specified as below.

- 4.4 Transbronchial mediastinal cryobiopsy after EBUS-TBNA
- 4.4.1 Opening of a window on the airway wall

The target lesion is supervised by ultrasound, and a high-frequency electric needle knife (Olympus KD-31C-1, Olympus, Tokyo, Japan) is inserted through the working channel of the EBUS bronchoscope, and an incision is then made (about 2 - 3 mm) on the airway wall adjacent to the target lesions. The knife is then advanced into the lesion under real-time ultrasound visualization, avoiding areas with abundant blood flow or massive necrosis. After

being confirmed within the lesion and the measurement of its insertion depth, the needle knife

is then withdrawn. The time from the insertion of the needle knife into the bronchoscope to its

removal from the work channel is recorded as the window-opening duration.

4.4.2 Cryobiopsy

An Erbe frozen probe (Erbe 20402-401, 1.1 mm, Erbe, Tübingen, Germany) is then

passed through the working channel of the EBUS bronchoscope, and advanced through the

window on the airway wall into the lesion under real-time ultrasound visualization, avoiding

areas with abundant blood flow or massive necrosis. After measuring the insertion depth of

the cryoprobe, the probe is activated to cool down with nitrous oxide for around 7 seconds.

Then the bronchoscopist gently extracts the cryoprobe tip with the rapidly frozen biopsy

specimen attached to it, and then withdraws the bronchoscope and the cryoprobe. The frozen

specimen is released from the cryoprobe by thawing in saline and it is then fixed in formalin.

4.4.3 One-time cryobiopsy is performed. Cryobiopsy time is recorded from the insertion

of the cryoprobe into the bronchoscope to its final exit from the working channel. The size of

each specimen is measured and recorded by its long axis and area.

4.5 Postbiopsy

Hemorrhage within the airway is assessed through the bronchoscope, especially in the

biopsy site. The procoagulants are locally used when necessary. Record all the

procedure-associated adverse events during the procedure, including bleeding, severe

hypoxemia, cardiac arrhythmia, hypotension, etc. The overall procedure duration is measured

from the insertion of bronchoscope to its removal from the patient's nose or mouth.

4.6 Procedure interruption

The EBUS procedure will be interrupted accordingly in the following situations:

7

1) Patients are intolerant to the bronchoscopic procedure;

2) The ultrasound fails to detect the lesion within 20 minutes;

3) The blood supply is so abundant in the lesion that is considered inappropriate to

continue biopsy due to the high risk;

4) The ultrasound identifies that the lesion is a cyst or abscess;

5) Severe adverse events occur during operation, such as severe bleeding. Bleeding is

classified as follows: grade 0, traces of blood not requiring suctioning; grade 1, bleeding only

requiring suctioning and hemostatic wedging for up to 2 minutes (two 1-minute cycles); grade

2, bleeding requiring hemostatic wedging for 3 minutes or more; grade 3, bleeding requiring

topical instillation of epinephrine or ice cold saline; and grade 4, bleeding requiring

hemodynamic support, transfusion of blood products, selective mainstem intubation,

bronchial blocker, hospital admission, or surgical intervention<sup>11, 12</sup>.

4.7 Histological assessment

All the specimens obtained from patients are sent to the Department of Pathology and

appropriately processed. The pathologic evaluation is made by the pathologists at each of the

centres, who are unaware of the patient recruitment for a clinical trial. In our study, the

pathological diagnosis is performed following the local workflow. All specimens are examined

by two pathologists.

4.8 Patient follow-up

Immediately after the operation, the patients are inquired about whether there are any

discomforts, and it is recorded if there are any. Chest X-ray or other imaging examinations are

performed within 24 hours to detect whether there is pneumothorax, pneumomediastinum, or

mediastinitis. Twenty-four hours after operation, a follow-up is conducted and the symptoms

are recorded, including fever, coughing, hemoptysis, chest pain, dyspnea, and so on.

Perioperative severe adverse events include moderate-to-severe bleeding (grade 3 or 4),

oversedation requiring ventilatory support or sedation reversal, pneumothorax with persistent

air leakage (> 5 days), unplanned hospital readmission, and death. ICU transfer within 48

hours after the procedure is also considered a severe adverse event. One month later, a second follow-up is conducted, and examinations such as X-ray or CT scan would be arranged according to patient symptom. The complications relative to the operation are recorded. Patients with an indefinite diagnosis (especially for benign disorders) are followed up continuously or receive surgical procedures (such as mediastinoscopy or surgical lymph node dissection), and the final diagnosis should be revised at any time if more reliable evidence supports new diagnosis. Six months later, imaging reexaminations are required for

patients with an indefinite diagnosis (especially for benign disorders).

### 5. Study endpoints

The co-primary outcomes are the diagnostic yield and safety of the EBUS procedure. The diagnostic yield of the EBUS procedure is defined as the percentage of patients for whom the EBUS procedures provided a definite diagnosis. Suspicious findings from the biopsy procedures are regarded as negative cases. Safety is evaluated with regard to the prevalence of the procedure-related adverse events.

Secondary end-points include the diagnostic yield of transbronchial mediastinal cryobiopsy, specimen adequacy and size, suitability of samples for molecular genetic assay, and duration of the bronchoscopic procedure.

#### 6. Data analysis

The full analysis set, including all the patients who do not violate the inclusion criteria and have undergone the biopsy, is used for demographic summaries and safety analyses. Inter-individual diagnostic analyses are performed based on the full analysis set, and the intra-individual diagnostic analyses include subjects receiving both EBUS-TBNA and mediastinal cryobiopsy, which are performed in concern of the potential intergroup differences<sup>13</sup>. Subgroup analyses are performed on disease etiology. Analyses of the

secondary outcomes are done in the combined biopsy population, except the analysis of

procedural duration that is based on the full analysis set.

Statistical analyses are performed using IBM SPSS 21.0 software (IBM Corp., Armonk,

NY, USA). Categorical variables are reported as counts and percentages, and continuous

variables as means and standard deviation. Pearson's Chi-squared or Fisher's exact test is

used to compare proportions, as appropriate. For continuous data, between-group

comparisons are performed by Student's t test or the Mann-Whitney U-test for parametric or

non-parametric data, respectively. A P<0.05 is considered to denote statistical significance.

Because of discussions within the research and statistical team about the need for more

details on how analyses are to be carried out, amendments to the data analysis section of the

protocol are made on Feb 8th 2022 before our analyses are started. The changes made are

that more specified information on the populations for the primary and subgroup analyses are

provided in this part.

7. Ethical considerations

The research group will ensure that this study is conducted in accordance with the

principles of the Declaration of Helsinki and Good Clinical Practice. All participants will be

asked to provide informed consent.

8. Risks and benefits

Similar to the application of standard needle aspiration biopsy, bleeding may occur during

the combined mediastinal sampling. In most situations, it requires no additional interventions.

Other adverse events include pneumothorax, infection, and hematoma or emphysema in

mediastinum; however, these occurrences are much less frequent<sup>7</sup>. The bronchoscopist will

try the best to operate carefully to avoid the damage to blood vessels and other important

tissues and organs. Patients will be reexamined by Chest X-ray or other imaging

10

examinations within 24 hours to detect whether there is pneumothorax, or emphysema,

hematoma, or infection in mediastinum.

Compared with the routine application of EBUS-TBNA alone, the operative duration of

the combined sampling may be prolonged by approximately 5 minutes (the duration required

for cryobiopsy), which may increase the discomfort of the patients. During the procedure,

conscious sedation, local anesthesia, and continuous vital signs and oxygen saturation

monitoring will be used to minimize the discomfort and ensure the safety of the patients.

Compared with the traditional EBUS-TBNA, the operation scheme of the combined

approach helps to obtain more intact tissues and improve diagnostic utilities. This lessened

the need for more invasive examinations and surgical procedures.

9. Privacy and personal information protection

The research group hereby promises to protect the privacy and personal information of

the subjects that participate in the study. The security measures for protecting the privacy and

confidentiality of personal information include hiding information that can identify the subjects

during data reports, restricting access to such information, data anonymity, and so on.

Legally, there are exceptions for researchers to protect the privacy and personal

information of subjects when inspections are required by administrative authorities, or ethics

committee, etc.

10. Funding

The study is funded by National Natural Science Foundation of China.

11. Reference

1. Wallace MB, Pascual JM, Raimondo M, et al. Minimally invasive endoscopic staging

11

of suspected lung cancer. JAMA 2008;299:540-6.

- 2. The American Thoracic Society and The European Respiratory Society. Pretreatment evaluation of non-small-cell lung cancer. Am J Respir Crit Care Med 1997;156:320-32.
- 3. Detterbeck FC, Jantz MA, Wallace M, Vansteenkiste J, Silvestri GA; American College of Chest Physicians. Invasive mediastinal staging of lung cancer: ACCP evidence-based clinical practice guidelines (2nd edition). Chest 2007;132:202S-220S.
- 4. Eapen GA, Shah AM, Lei X, et al. Complications, consequences, and practice patterns of endobronchial ultrasound-guided transbronchial needle aspiration: Results of the AQuIRE registry. Chest 2013;143:1044-53.
- 5. Franke KJ, Bruckner C, Szyrach M, Ruhle KH, Nilius G, Theegarten D. The contribution of endobronchial ultrasound-guided forceps biopsy in the diagnostic workup of unexplained mediastinal and hilar lymphadenopathy. Lung 2012;190:227-32.
- 6. Zhang J, Fu WL, Huang ZS, et al. Primary Mediastinal Seminoma Achieved by Transbronchial Mediastinal Cryobiopsy. Respiration 2020;99:426-30.
- 7. Zhang J, Guo JR, Huang ZS, et al. Transbronchial mediastinal cryobiopsy in the diagnosis of mediastinal lesions: a randomised trial. Eur Respir J 2021;58:2100055.
- 8. Nakajima T, Anayama T, Koike T, et al. Endobronchial ultrasound doppler image features correlate with mRNA expression of HIF1-α and VEGF-C in patients with non-small-cell lung cancer. J Thorac Oncol 2012;7:1661-7.
- 9. Nakajima T, Anayama T, Shingyoji M, Kimura H, Yoshino I, Yasufuku K. Vascular image patterns of lymph nodes for the prediction of metastatic disease during EBUS-TBNA for mediastinal staging of lung cancer. J Thorac Oncol 2012;7:1009-14.
- 10. Wahidi MM, Herth F, Yasufuku K, et al. Technical Aspects of Endobronchial Ultrasound-Guided Transbronchial Needle Aspiration: CHEST Guideline and Expert Panel Report. Chest. 2016;149(3):816-35.
- 11. Yarmus L, Akulian J, Gilbert C, et al. Cryoprobe transbronchial lung biopsy in patients after lung transplantation: a pilot safety study. Chest 2013;143:621-6.
  - 12. Du Rand IA, Blaikley J, Booton R, et al. British Thoracic Society guideline for

diagnostic flexible bronchoscopy in adults: accredited by NICE. Thorax 2013;68:i1-i44.

13. Takwoingi Y, Leeflang MM, Deeks JJ. Empirical evidence of the importance of comparative studies of diagnostic test accuracy. Ann Intern Med 2013;158:544-54.